CLINICAL TRIAL: NCT04595370
Title: A Phase 2b, Randomised, Double-Blind, Active Controlled, Multi Centre Study to Evaluate the Efficacy, Safety and Tolerability of Oral AZD9977 and Dapagliflozin Treatment in Patients With Heart Failure and Chronic Kidney Disease
Brief Title: Efficacy, Safety and Tolerability of AZD9977 and Dapagliflozin in Participants With Heart Failure and Chronic Kidney Disease
Acronym: MIRACLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6402C00001; 2020-003126-23 (EudraCT Number)
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Chronic Kidney Disease
Keywords: Heart Failure; Type 2 diabetes mellitus; Diabetic kidney disease; Chronic kidney disease; Mineralocorticoid receptor modulator; Sodium-glucose co-transporter-2 inhibitor; AZD9977; Dapagliflozin; Urinary albumin creatinine ratio
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — AZD9977; dapagliflozin

STUDY DESIGN:
Intervention Model Description: Participants who meet the eligibility criteria will be randomized to one of the following treatment group:
  1. AZD9977 Dose A + dapagliflozin 10 mg
  2. AZD9977 Dose B + dapagliflozin 10 mg
  3. AZD9977 Dose C + dapagliflozin 10 mg
  4. Dapagliflozin 10 mg
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZD9977 Dose A + dapagliflozin 10 mg (Experimental): Participants will receive once daily oral dose A of AZD9977 and 10 mg dapagliflozin for 12 weeks.
  Interventions: Drug: AZD9977; Drug: Dapagliflozin
- AZD9977 Dose B + dapagliflozin 10 mg (Experimental): Participants will receive once daily oral dose B of AZD9977 and 10 mg dapagliflozin for 12 weeks.
  Interventions: Drug: AZD9977; Drug: Dapagliflozin
- AZD9977 Dose C + dapagliflozin 10 mg (Experimental): Participants will receive once daily oral dose C of AZD9977 and 10 mg dapagliflozin for 12 weeks.
  Interventions: Drug: AZD9977; Drug: Dapagliflozin
- Dapagliflozin 10 mg (Experimental): Participants will receive once daily oral dose of dapagliflozin 10 mg alone for 12 weeks.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: AZD9977 — Participants will receive AZD9977 as per the arms they are randomized.
  Arms: AZD9977 Dose A + dapagliflozin 10 mg; AZD9977 Dose B + dapagliflozin 10 mg; AZD9977 Dose C + dapagliflozin 10 mg
Drug: Dapagliflozin — Participants will receive dapagliflozin as per the arms they are randomized.

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of AZD9977 in combination with dapagliflozin compared with dapagliflozin alone and to assess the dose-response relationship, dapagliflozin alone and 3 doses of AZD9977 combined with dapagliflozin on urinary albumin to creatinine ratio (UACR). The study will be conducted in participants with heart failure (HF) with left ventricular ejection fraction (LVEF [below 60%]) and chronic kidney disease (CKD) with estimated glomerular filtration rate (eGFR [between ≥ 20 and ≤ 60 mL/min/1.73 m^2, with at least 20% of participants with eGFR ≥ 20 to <30 mL/min/1.73^2 and a maximum of 35% of participants with eGFR ≥ 45 mL/min/1.73 m^2]).

DETAILED DESCRIPTION:
After screening, eligible participants will undergo a run-in period where all participants receive dapagliflozin for up to 7 weeks depending on pre-study use of SGLT2i or not. At the end of the run-in period, eligible participants will be randomly assigned with a 1:1:1:1 ratio to receive once daily administration of one of the following 4 study treatments group for 12 weeks. To ensure blinding, the study treatment will be administered in the form of 3 oral capsules of AZD9977 or placebo and 1 oral tablet or dapagliflozin.

1. AZD9977 Dose A + dapagliflozin 10 mg
2. AZD9977 Dose B + dapagliflozin 10 mg
3. AZD9977 Dose C + dapagliflozin 10 mg
4. Dapagliflozin 10 mg

Participants will be randomized to one of the above treatment group, according to type 2 diabetes mellitus [T2DM (yes/no)] and eGFR (≥ 20 to <30 mL/min/1.73^2; or ≥ 30 to < 45 mL/min/1.73^2; or ≥45 mL/min/1.73^2).

The total duration of participation will be approximately 22 to 24weeks.

ELIGIBILITY:
Inclusion Criteria:

Participants are included in the study if any of the following criteria apply:

* Documented diagnosis of stable symptomatic HF (New York Heart Association class II-III) at screening, and a medical history of typical symptoms and signs of HF in those who are currently receiving loop diuretic treatment
* Left ventricular ejection fraction <60% documented by the most recent echocardiogram or cardiac magnetic resonance imaging within the last 12 months prior to screening
* Stable background treatment for HF, hypertension, diabetes mellitus or renal disease according to guidelines
* N-terminal-pro-brain natriuretic peptide (NT proBNP) ≥300 pg/mL for participants with sinus rhythm at screening; and NT proBNP ≥600 pg/mL for participants with atrial fibrillation/flutter at screening
* The eGFR ≥30 and ≤60 mL/min/1.73^2 (by CKD- EPI formula) and UACR ≥30 mg/g (3 mg/mmol) and <3000 mg/g (300 mg/mmol)
* Body mass index less than 40 kg/m^2
* Serum/plasma K+ level ≥ 3.5 and < 5.0 mmol/L within 10 days prior to randomization
* Serum/ plasma Na+ level within normal reference values within 10 days prior to randomization
* Systolic blood pressure should be at protocol defined range at randomization (Visit 3), with no change to antihypertensive treatments in previous 3 weeks
* Male or female of non-childbearing potential
* All participants must follow protocol defined contraceptives procedures

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Primary glomerulopathy, vasculitic renal disease, prior dialysis or unstable rapidly progressing renal disease, autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis or anti-neutrophil cytoplasm antibody-associated vasculitis
* Participants with currently decompensated HF requiring hospitalization for optimization of HF treatment and are not on stable HF therapy at the time of enrollment
* HF due to cardiomyopathies
* High output HF (e.g., due to hyperthyroidism or Paget's disease)
* HF due to pericardial disease, congenital heart disease or clinically significant uncorrected primary cardiac valvular disease or planned cardiac valve repair/replacement
* Participants with uncontrolled diabetes mellitus (Glycated hemoglobin >10%)
* Participants with Type 1 diabetes mellitus
* Intermittent or persistent 2nd or 3rd degree atrioventricular block, sinus node dysfunction with clinically significant bradycardia or sinus pauses, not treated with a pacemaker
* History of any life-threatening cardiac dysrhythmia or uncontrolled ventricular rate in participants with atrial fibrillation or atrial flutter
* Acute coronary syndrome and/or elective/non-elective percutaneous cardiac interventions (within 3 months) prior to randomisation or is planned to undergo any of these procedures during the study
* Any major cardiovascular (eg, open chest, coronary artery bypass grafting or valvular repair/replacement) or major non-cardiovascular surgery within 3 months prior to randomisation or is planned to undergo any cardiovascular surgery during the study
* Heart transplantation or left ventricular assist device at any time or if these are planned
* Kidney or any organ transplantation or if these are planned
* Medical conditions associated with development of hyperkalaemia (Addison's disease )
* History or ongoing allergy/hypersensitivity, to sodium-glucose co-transporter-2 inhibitor (SGLT2i e.g., dapagliflozin, empagliflozin)
* Stroke, transient ischemic attack, carotid surgery, or carotid angioplasty within previous 3 months prior to randomisation
* Hepatic disease, including hepatitis and/or hepatic impairment (Child-Pugh class A-C), and aspartate aminotransferase or alanine transaminase or total bilirubin should be in protocol defined range at time of screening and/ or within 7 days prior to randomization
* Participants with newly detected pathological laboratory values or an ongoing disease condition
* If the participants clinical signs and symptoms consistent with COVID-19, and has been previously hospitalized with COVID-19 infection and did not fully recover their previous health status
* Previous randomization in the present study
* Prior medical treatment with an mineralocorticoid receptor antagonist where the medication was taken within 90 days prior to screening
* Current or prior treatment within 6 months prior to screening with cytotoxic therapy, immunosuppressive therapy, or other immunotherapy

Ages: 21 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McMurray, Principal Investigator — University of Glasgow, United Kingdom
Locations (128):
- United States (25):
  - Research Site, Beverly Hills, California
  - Research Site, Fountain Valley, California
  - Research Site, Northridge, California
  - Research Site, South Gate, California
  - Research Site, Hialeah, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Methuen, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, The Bronx, New York
  - Research Site, New Bern, North Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sherman, Texas
  - Research Site, Webster, Texas
- Research Site, Roeselare, Belgium
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
- Canada (4):
  - Research Site, Peterborough, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (3):
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Uherské Hradiště
- Denmark (3):
  - Research Site, Aarhus
  - Research Site, Herlev
  - Research Site, Svendborg
- Germany (4):
  - Research Site, Dresden
  - Research Site, Frankfurt
  - Research Site, Jena
  - Research Site, Leipzig
- Hungary (5):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Miskolc
  - Research Site, Orosháza
- India (4):
  - Research Site, Ahmedabad
  - Research Site, Chennai
  - Research Site, Kolkata
  - Research Site, Pune
- Research Site, Roma, Italy
- Japan (19):
  - Research Site, Chūōku
  - Research Site, Hamada-shi
  - Research Site, Hamamatsu
  - Research Site, Hanyu-shi
  - Research Site, Itabashi-ku
  - Research Site, Kasugai-shi
  - Research Site, Kawaguchi
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Matsudo-Shi
  - Research Site, Matsumoto-shi
  - Research Site, Ono
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Takasago-shi
  - Research Site, Takasaki-shi
  - Research Site, Ueda-shi
  - Research Site, Yokohama
- Lithuania (4):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Šiauliai
  - Research Site, Vilnius
- Poland (14):
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Oświęcim
  - Research Site, Oława
  - Research Site, Pabianice
  - Research Site, Poznan
  - Research Site, Skorzewo
  - Research Site, Sopot
  - Research Site, Szczecin
  - Research Site, Torun
  - Research Site, Warsaw
- Russia (5):
  - Research Site, Kazan'
  - Research Site, Kazan, Tatarstan
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Slovakia (6):
  - Research Site, Banská Bystrica
  - Research Site, Brezno
  - Research Site, Lučenec
  - Research Site, Prešov
  - Research Site, Svidník
  - Research Site, Trenčín
- South Korea (4):
  - Research Site, Busan
  - Research Site, Gangwon-do
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, El Palmar
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Chaingmai
  - Research Site, Khon Kaen
- Turkey (Türkiye) (2):
  - Research Site, Adana
  - Research Site, Kocaeli
- Ukraine (3):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis_D6402C00001 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6402C00001&attachmentIdentifier=fddab4bc-57ea-45ba-b963-ae71d1eb0839&fileName=Redacted_CSR_Synopsis_D6402C00001.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 26-January-2021 (first subject first visit) to 22-September-2023 (last subject last visit).
Pre-assignment Details: Participants who signed the Informed Consent Form (ICF) were enrolled into study. The study included an optional pre-screening visit.
Groups:
- AZD9977 15 mg + Dapagliflozin 10 mg: Participants received AZD9977 15 mg and dapagliflozin 10 mg orally once daily for 12 weeks.
- AZD9977 50 mg + Dapagliflozin 10 mg: Participants received AZD9977 50 mg and dapagliflozin 10 mg orally once daily for 12 weeks.
- AZD9977 150 mg + Dapagliflozin 10 mg: Participants received AZD9977 150 mg and dapagliflozin 10 mg orally once daily for 12 weeks.
- AZD9977 150 mg: Participants received AZD9977 150 mg and placebo matching to dapagliflozin orally once daily for 12 weeks.
- Dapagliflozin 10 mg: Participants received dapagliflozin 10 mg and placebo matching to AZD9977 orally once daily for 12 weeks.
- Placebo: Placebo participants received placebo matching to AZD9977 and dapagliflozin orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo
Started | 35 | 33 | 36 | 7 | 35 | 7
Completed | 33 | 25 | 27 | 6 | 29 | 6
Not Completed | 2 | 8 | 9 | 1 | 6 | 1
Not completed — Subjects randomised, not treated, Protocol Deviation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Subjects randomised, not treated, Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 3 | 1 | 1 | 1
Not completed — Withdrawal of Consent | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Protocol-Specified Withdrawal Criterion Met | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participants discontinued study treatment due to other reasons | 0 | 2 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Total 153 participants were randomized but 9 participants were excluded from full analysis set (FAS) due to good clinical practice (GCP) misconduct at site. Hence, 144 participants were included in FAS.
  FAS included all participants who were randomized and either received or did not receive any study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo | Total
Number analyzed (Participants) | 34 | 31 | 35 | 6 | 33 | 5 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (7.1) | 72.4 (8.4) | 73.7 (8.1) | 77.0 (8.7) | 72.2 (9.4) | 77.2 (5.8) | 72.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 8 | 1 | 10 | 1 | 36
  Male | 23 | 26 | 27 | 5 | 23 | 4 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 3 | 7 | 0 | 3 | 0 | 17
  Black or African American | 0 | 1 | 1 | 0 | 2 | 1 | 5
  White | 30 | 27 | 27 | 6 | 28 | 4 | 122

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Urinary Albumin to Creatinine Ratio (UACR) at Week 12
Description: The effect of AZD9977 in combination with dapagliflozin compared with dapagliflozin alone on UACR assessed. Urine samples were collected for the analysis of UACR. UACR (milligrams per gram [mg/g]) was calculated as 10 x urine albumin (mg per deciliter [mg/dL])/urine creatinine (g/dL). Change from baseline in UACR at the end of 12 weeks of study treatment was calculated as the average of the UACR values at Week 12 and was analyzed by a mixed-effects model for repeated measures (MMRM). Due to early removal of arms (AZD9977 150 mg monotherapy and Placebo), the study objectives were revised and the MMRM analysis included the 4 remaining arms (AZD9977 15 mg + Dapagliflozin, AZD9977 50 mg + Dapagliflozin, AZD9977 150 mg + Dapagliflozin, and Dapagliflozin 10 mg). Since 2 arms were removed from the study resulting in fewer participants only descriptive statistics are shown for those two arms without formal comparison.
Time Frame: Baseline (Day 1) to Week 12
Population: Full analysis set included all participants who were randomized and either received or did not receive any study intervention. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 32 | 23 | 25 | 5 | 28 | 3
Percent change from baseline | -56.391 [-71.528 to -33.207] | -42.085 [-64.174 to -6.376] | -58.047 [-73.560 to -33.430] | -45.01 [NA to NA] — NA indicates that the lower and upper limits of the 95% CI were not calculated due to insufficient number of participants enrolled in this arm. | -34.318 [-58.204 to 3.220] | 230.32 [NA to NA] — NA indicates that the lower and upper limits of the 95% CI were not calculated due to insufficient number of participants enrolled in this arm.
Statistical Analysis 1: Comparison: AZD9977 15 mg + Dapagliflozin 10 mg vs AZD9977 50 mg + Dapagliflozin 10 mg vs AZD9977 150 mg + Dapagliflozin 10 mg vs Dapagliflozin 10 mg; Test type: Other; p = 0.3645, F-Test; F test statistics = 1.07

2. Secondary Outcome: Percent Change From Baseline in Urinary Albumin to Creatinine Ratio (UACR) at 12 Weeks to Assess Dose-Response Relationship
Description: The dose-response relationship of dapagliflozin alone and 3 doses of AZD9977 combined with dapagliflozin on UACR was assessed. Urine samples were collected for the analysis of UACR. UACR (mg/g) was calculated as 10 x urine albumin (mg/dL)/urine creatinine (g/dL). Change from baseline in UACR at the end of 12 weeks of study treatment was calculated as the average of the UACR values at Week 12 and was analyzed by a mixed-effects model for repeated measures (MMRM). Due to early removal of arms (AZD9977 150 mg monotherapy and Placebo), the study objectives were revised and the MMRM analysis included the 4 remaining arms (AZD9977 15 mg + Dapagliflozin, AZD9977 50 mg + Dapagliflozin, AZD9977 150 mg + Dapagliflozin, and Dapagliflozin 10 mg). Since 2 arms were removed from the study resulting in fewer participants, only descriptive statistics was shown for those two arms without formal comparison.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 32 | 23 | 25 | 5 | 28 | 7
Percent change from baseline | -56.391 [-71.528 to -33.207] | -42.085 [-64.174 to -6.376] | -58.047 [-73.560 to -33.430] | -45.01 [NA to NA] — NA indicates that the lower and upper limits of the 95% CI were not calculated due to insufficient number of participants enrolled in this arm. | -34.318 [-58.204 to 3.220] | 230.32 [NA to NA] — NA indicates that the lower and upper limits of the 95% CI were not calculated due to insufficient number of participants enrolled in this arm.
Statistical Analysis 1: Comparison: AZD9977 15 mg + Dapagliflozin 10 mg vs Dapagliflozin 10 mg; Test type: Other; p = 0.1588, Mixed Models Analysis; Percent difference between treatment = -33.606, 95% CI 2-sided [-62.530 to 17.644]
Statistical Analysis 2: Comparison: AZD9977 50 mg + Dapagliflozin 10 mg vs Dapagliflozin 10 mg; Test type: Other; p = 0.6846, Mixed Models Analysis; Percent difference between treatment = -11.826, 95% CI 2-sided [-52.195 to 62.634]
Statistical Analysis 3: Comparison: AZD9977 150 mg + Dapagliflozin 10 mg vs Dapagliflozin 10 mg; Test type: Other; p = 0.1398, Mixed Models Analysis; Percent difference between treatment = -36.127, 95% CI 2-sided [-64.850 to 16.066]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The safety and tolerability of AZD9977 combined with dapagliflozin 10 mg, AZD9977 monotherapy, dapagliflozin 10 mg monotherapy and placebo was assessed.
Time Frame: From baseline (Day 1) until Day 113
Population: Safety analysis set included all participants who were randomized and received any study intervention. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 33 | 31 | 34 | 6 | 33 | 5
Participants
  Any AE | 9 | 12 | 18 | 5 | 14 | 3
  Any SAE | 1 | 3 | 2 | 0 | 4 | 2
  Any SAE with outcome death | 0 | 2 | 0 | 0 | 1 | 0
  Any AE leading to discontinuation of IP | 0 | 4 | 3 | 1 | 1 | 1
  Any AE leading to withdrawal from study | 0 | 5 | 2 | 0 | 1 | 0
  Any AE leading to dose interruption | 1 | 1 | 1 | 0 | 3 | 1

4. Secondary Outcome: Change From Baseline in Serum Potassium (K+)
Description: Effect of AZD9977 combined with dapagliflozin 10 mg, AZD9977 monotherapy, dapagliflozin 10 mg monotherapy and placebo on serum K+ was assessed.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 27 | 21 | 25 | 4 | 25 | 3
millimoles per liter (mmol/L) | 0.056 [-0.106 to 0.219] | 0.003 [-0.184 to 0.190] | 0.109 [-0.061 to 0.279] | 0.55 [NA to NA] — NA indicates that the lower and upper limits of the 95% CI were not calculated due to insufficient number of participants enrolled in this arm. | 0.040 [-0.129 to 0.209] | 0.03 [NA to NA] — NA indicates that the lower and upper limits of the 95% CI were not calculated due to insufficient number of participants enrolled in this arm.

5. Secondary Outcome: Absolute Value of Serum Potassium Over Time
Description: as for outcome 4
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 30 | 25 | 29 | 5 | 33 | 5
mmol/L
  Baseline | 4.60 (0.38) | 4.44 (0.61) | 4.46 (0.44) | 4.50 (0.38) | 4.60 (0.66) | 4.50 (0.28)
  Week 12: number analyzed (Participants) | 27 | 21 | 25 | 4 | 25 | 3
  Week 12 | 4.62 (0.50) | 4.53 (0.43) | 4.63 (0.43) | 5.00 (0.61) | 4.64 (0.40) | 4.33 (0.32)

6. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: Effect of AZD9977 combined with dapagliflozin 10 mg, AZD9977 monotherapy, dapagliflozin 10 mg monotherapy and placebo on eGFR was assessed.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 26 | 21 | 24 | 4 | 23 | 3
mL/min/1.73 m^2 | -1.432 [-4.305 to 1.441] | -1.160 [-4.351 to 2.030] | -5.307 [-8.295 to -2.320] | -0.923 [NA to NA] — NA indicates that the lower and upper limits of the 95% CI were not calculated due to insufficient number of participants enrolled in this arm. | -3.498 [-6.528 to -0.469] | 6.880 [NA to NA] — NA indicates that the lower and upper limits of the 95% CI were not calculated due to insufficient number of participants enrolled in this arm.

7. Secondary Outcome: Absolute Value of eGFR Over Time
Description: Effect of all doses of AZD9977 combined with dapagliflozin 10 mg, AZD9977 monotherapy, dapagliflozin 10 mg monotherapy and placebo on eGFR was assessed
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 32 | 31 | 33 | 5 | 32 | 5
mL/min/1.73 m^2
  Baseline | 41.341 (12.902) | 38.586 (10.155) | 43.663 (16.168) | 36.874 (12.626) | 41.895 (12.791) | 40.288 (15.176)
  Week 12: number analyzed (Participants) | 26 | 21 | 24 | 4 | 23 | 3
  Week 12 | 41.219 (15.112) | 39.429 (8.998) | 39.063 (13.819) | 34.075 (21.071) | 37.973 (11.571) | 48.920 (21.111)

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) until Day 113
Description: Safety set included all participants who were randomized and received any study intervention.
  All AEs that were reported with an onset date and time, or worsening, on or after date and time of first dose of IP up to and including 28 days after last dose of IP were included in the safety analysis.
Arm/Group | AZD9977 15 mg + Dapagliflozin 10 mg | AZD9977 50 mg + Dapagliflozin 10 mg | AZD9977 150 mg + Dapagliflozin 10 mg | AZD9977 150 mg | Dapagliflozin 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 2/31 | 0/34 | 0/6 | 1/33 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/33 | 3/31 | 2/34 | 0/6 | 4/33 | 2/5
Other Adverse Events (participants affected / at risk) | 1/33 | 4/31 | 13/34 | 5/6 | 7/33 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9977 15 mg + Dapagliflozin 10 mg (N=33) | AZD9977 50 mg + Dapagliflozin 10 mg (N=31) | AZD9977 150 mg + Dapagliflozin 10 mg (N=34) | AZD9977 150 mg (N=6) | Dapagliflozin 10 mg (N=33) | Placebo (N=5)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9977 15 mg + Dapagliflozin 10 mg (N=33) | AZD9977 50 mg + Dapagliflozin 10 mg (N=31) | AZD9977 150 mg + Dapagliflozin 10 mg (N=34) | AZD9977 150 mg (N=6) | Dapagliflozin 10 mg (N=33) | Placebo (N=5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrolment stopped early because of slow recruitment. Therefore, pre-specified sample size of 500 and planned statistical power were not achieved. Nine subjects were excluded from analysis due to site misconduct and GCP non-compliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (2):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT04595370/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT04595370/SAP_001.pdf